CLINICAL TRIAL: NCT03240666
Title: Multicentric Clinical Trials on the Prevalence of Entamoeba Gingivalis and Its Associated Bacterial Flora in Patients With Periodontitis
Brief Title: Protozoans in Biofilm From Patients With Periodontitis
Acronym: Paro-Proto
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016/PARO-PROTO-BISSON/ER
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2020-07

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Bacterial DNA, protozoan DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non applicable — non applicable

SUMMARY:
The buccal cavity is colonized by numerous microorganisms whose the number and composition could be modified with medical background (diseases and drugs) and the level of oral hygiene of the patients. Among all microorganisms identified in the periodontium, few of them are implicated in the etiopathogenesis of periodontal pathologies. To date, four major bacteria are identified for their ability to degrade periodontal tissues.

Although the periodontitis is established to be the consequence of bacterial virulence and immune dysfunction, these factors fail to explain the refractory periodontitis of some patients to etiologic treatment .

Others microorganisms such as protozoans could have an impact on this disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years-old
* consulting in periodontal department of CHRU
* Patients with moderate to severe periodontitis
* At least 2 periodontal sites with PPD ≥ 5mm and one healthy site
* No scaling root planing in the last 6 months
* Patients insured under the Franch social security system

Exclusion Criteria:

* Pregnants patients
* Patients with antibiotic therapy and/ or all medecines which could modify the buccal microbiota in the last 6 months
* Tooth with endodontics periapical lesion
* Patients having a scaling root planing in the last 6 months
* Patients with guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients consulting to periodontal department of CHRU (Nancy-Nice- Toulouse) presenting at least two PPD of 5mm and more, without any medecines which could modify microbiota were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 231 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
presence of protozoans | 6 months after the last inclusion: DNA samples were frozen and identified later.
  identification of protozoans by molecular technique (PCR) -

SECONDARY OUTCOMES:
Periodontal pocket depth (PPD in mm) | One day: measure realised during examination of the patient for periodontal treatment.
  Measure of PPD thanks to periodontal probe
Clinical attachment Loss (CAL in mm) | One day: measure realied during clincal examination of patient.
  Measure of CAL with periodontal probe
Plaque and gingival index | One day: measure of index during the clinical examination of patient.
  Measure of plaque and gingival index (Loe and Silness, Silness and Loe)
Mobility of tooth | One day: measure of tooth mobility during the clinical examination of patient.
  Measure of tooth mobility: Yes or not
Bleeding On Probing (BOP) | One day: measure of BOP during the clinical examination of patient.
  Measure of BOP : Yes or not

CONTACTS AND LOCATIONS:
Locations (1):
- Catherine BISSON, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided
non applicable